CLINICAL TRIAL: NCT00349401
Title: Intrathecal Ketorolac in Patients With Intrathecal Morphine Dose Escalation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated. No subjects were screened or enrolled.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: P01NS041386_TRIAL3; P01NS041386 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2009-05

CONDITIONS: Pain
Keywords: pain; chronic pain; morphine; ketorolac
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Ketorolac; Morphine

INTERVENTIONS:
Drug: ketorolac
Drug: morphine

SUMMARY:
The purpose of this study is to determine how the drug ketorolac, when given with the spinal morphine, affects pain.

DETAILED DESCRIPTION:
This study is part of a pain center grant that focuses on how pain, especially chronic neuropathic pain, alters the response to traditional and non-traditional analgesics (pain medications).

To treat persons with chronic pain, doctors sometimes implant a permanent tube in the spinal space in the back to give pain medicines. This tube, also called a spinal pump, is used to administer pain medicine directly to the spinal space. The most commonly used medicine given through the spinal pump is morphine which works well for most people, but sometimes loses tolerance, and larger and larger doses are needed, causing many side effects.

The purpose of this study is to find out if another medicine, ketorolac, when given with morphine in the spinal space, can stop or reverse the need for larger and larger doses of morphine. In animals, ketorolac has been shown to slow the need for an increase in morphine dosage and to reduce the morphine dose, while giving good pain control.

This study will enroll 30 individuals with chronic pain below the chest, caused by nerve injury, who are receiving morphine through a spinal pump. After learning to estimate pain accurately using thermal heat testing, participants will be randomly assigned to one of two study groups. Group one will receive the active study medication, ketorolac, while group two receives an inactive control (placebo). All participants will receive morphine (administered through the spinal pump). Afterwards, participants will rate their levels of pain, and provide samples of their spinal fluid (taken from the spinal tube/pump) for study. The above procedure will be repeated over a 4-week period.

Duration of the study for participants is 4 weeks, and includes ten visits to the research center, each lasting less than one hour.

ELIGIBILITY:
Inclusion Criteria:

* Implanted spinal pump for at last 9 months
* Must be receiving and the dose must have been doubled in the past 6 months
* Currently taking 60-200 mg morphine equivalent as oral rescue per day
* Men and women, ages 18-70
* Weigh no more that 250 pounds
* Neuropathic pain

Exclusion Criteria:

* Pregnancy
* Unstable medical problems (heart lung, liver, kidney, or nervous system)
* Allergy to morphine, ketorolac, or drugs which may be used to treat side effects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12

PRIMARY OUTCOMES:
VAS pain.
Primary analysis will be the comparison between ketorolac and placebo groups.

SECONDARY OUTCOMES:
Change in oral opioid dose.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences; Richard Rauck, M.D., Principal Investigator — The Center for Clinical Research